CLINICAL TRIAL: NCT00000752
Title: Management of HIV-Infected Patients at Risk of Recurrent Purulent Sinusitis: Role of Anti-Inflammatory, Antibacterial, and Decongestant Prophylaxis
Brief Title: Preventing Frequent Sinus Infections in HIV-Infected Patients
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Adams Laboratories (Industry); Glaxo Wellcome (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: ACTG 186
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; Sinusitis
Keywords: Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; cefuroxime axetil; Beclomethasone; Guaiacol Glyceryl Ether; Sinusitis; Ephedrine
MeSH Terms: conditions — HIV Infections; Sinusitis; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Pseudoephedrine; Guaifenesin; cefuroxime axetil; Beclomethasone

INTERVENTIONS:
Drug: Pseudoephedrine hydrochloride
Drug: Guaifenesin
Drug: Cefuroxime axetil
Drug: Beclomethasone dipropionate

SUMMARY:
To evaluate the additional effectiveness of an anti-inflammatory nasal spray ( beclomethasone dipropionate ) and a broad spectrum antibiotic ( cefuroxime axetil ) over decongestant ( Deconsal II ) alone, when these agents are given individually or in combination for the prevention of recurrent paranasal sinus infection in patients with HIV infection. To compare the clinical utility of paranasal sinus radiographs with computed tomograms (CTs) in the evaluation and management of HIV-infected patients with recurrent paranasal sinus infection. To determine relevant prognostic factors and the microbiologic etiology of maxillary sinusitis in this patient population.

Sinusitis is common among HIV-infected patients and is likely to be recurrent or refractory to traditional therapy, particularly in patients with advanced immunosuppression. An intervention aimed at prevention of recurrent sinus disease in HIV-infected patients appears to be warranted.

DETAILED DESCRIPTION:
Sinusitis is common among HIV-infected patients and is likely to be recurrent or refractory to traditional therapy, particularly in patients with advanced immunosuppression. An intervention aimed at prevention of recurrent sinus disease in HIV-infected patients appears to be warranted.

Patients receive 21-42 days of antibiotic therapy for the defining episode of sinusitis. Following discontinuation of antibiotics, screening evaluations are performed. Within 7 days following completion of antibiotics, patients with clinical resolution begin 14 +/- 3 days of decongestant therapy with oral Deconsal II, a drug combining pseudoephedrine, a decongestant, and guaifenesin, an expectorant. Following decongestant therapy, patients undergo entry evaluations, including nasal endoscopy and sinus radiograph. Patients with continued clinical resolution and no purulence on endoscopy are then randomized to receive decongestant alone or in combination with nasal steroid (beclomethasone dipropionate) or antibiotic (cefuroxime axetil) or both. Treatment continues for a minimum of 52 weeks and a maximum of 104 weeks. Patients are followed at weeks 4, 8, and 12 and every 8 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Antiretroviral agents (both approved and investigational).
* Biologic response modifiers.
* Systemic chemotherapy.
* Chemoprophylaxis for Pneumocystis carinii pneumonia (PCP), candidiasis, and herpes.
* Adjuvant systemic corticosteroids with appropriate antibiotic therapy for moderate to severe PCP.
* Maintenance therapy with pyrimethamine, sulfadiazine, amphotericin B, fluconazole, ketoconazole, or acyclovir.
* Treatment with ganciclovir, foscarnet, or antimycobacterial drugs for CMV disease or mycobacterial infections.
* Non-beta lactam antibacterial agents for other infections (beta lactam antibacterial agents are allowed if study drugs are temporarily discontinued).
* Antihistamines and saline nasal sprays.

Concurrent Treatment:

Allowed:

* Radiation therapy.

Patients must have:

* HIV infection.
* At least one episode of symptomatic maxillary sinusitis, with clinical resolution following antibiotic therapy.
* Life expectancy of at least 12 months.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Concurrent infection caused by cytomegalovirus or Mycobacterium avium Complex.
* Significant emotional disorder or psychosis.
* Conditions such as dementia that would substantially impair study compliance.
* Evidence of significant malabsorption, ileus, or significant emesis that would inhibit drug absorption.
* Inability to tolerate a minimum administration of one tablet of oral Deconsal II daily.

Concurrent Medication:

Excluded:

* Prescription or over-the-counter nasal steroids, decongestants, or topical vasoconstrictors (ephedrine, oxymetazoline).

Patients with the following prior condition are excluded:

* History of an acute hypersensitivity reaction to any penicillin or cephalosporin, characterized by urticaria, hypotension, or laryngeal edema.

Active substance abuse that would impair study compliance.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Study Completion 1993-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J Zurlo, Study Chair; JA McCutchan, Study Chair
Locations (10):
- United States (10):
  - Univ of California / San Diego Treatment Ctr, San Diego, California
  - Stanford at Kaiser / Kaiser Permanente Med Ctr, San Francisco, California
  - Montefiore Drug Treatment Ctr / Bronx Municipal Hosp, The Bronx, New York
  - Montefiore Family Health Ctr / Bronx Municipal Hosp, The Bronx, New York
  - Samaritan Village Inc / Bronx Municipal Hosp, The Bronx, New York
  - Jack Weiler Hosp / Bronx Municipal Hosp, The Bronx, New York
  - Montefiore Med Ctr / Bronx Municipal Hosp, The Bronx, New York
  - Montefiore Med Ctr Adolescent AIDS Program, The Bronx, New York
  - North Central Bronx Hosp / Bronx Municipal Hosp, The Bronx, New York
  - Thomas Jefferson Univ Hosp, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Zurlo JJ, Feuerstein IM, Lebovics R, Lane HC. Sinusitis in HIV-1 infection. Am J Med. 1992 Aug;93(2):157-62. doi: 10.1016/0002-9343(92)90045-d. PMID 1353944